CLINICAL TRIAL: NCT05737979
Title: Modified Rekovelle and Menopur Combination Protocol to Avoid Monitoring Before Day 10 of Stimulation
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: 3189
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Infertility; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women undergoing IVF: Women undergoing an antagonist in vitro fertilization cycle using Rekovelle and Menopur for stimulation
  Interventions: Other: Study chart review

INTERVENTIONS:
Other: Study chart review — Evaluation of the IVF cycle using the prescribed medication

SUMMARY:
Follitropin delta (Rekovelle) algorithm established by Ferring provides personalized gonadotrophin doses based on each patient's weight and AMH. As a result, risks of stimulation failure or ovarian hyperstimulation syndrome (OHSS) during an in vitro fertilization (IVF) cycle are minimized.

As a standard practice for OHSS prevention at clinique ovo, women undergoing IVF will have a scheduled ultrasound and blood test on the sixth day of their stimulation treatment. However, with the determination of the Rekovelle and Menopur algorithm, the risks of OHSS before the tenth day have been considerably minimized.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the necessity of programming an ultrasound and blood test prior to the tenth day of ovarian stimulation when women are on personalized doses of Rekovelle and Menopur duting an antagonist IVF cycle. Based on the results of the analysis, we will assess the economic impact that programming an ultrasound and blood test at day 10 might have.

ELIGIBILITY:
Inclusion Criteria:

* Women of 18 years of age or older having provided consent to chart access for scientific publication in the IVF consent form
* Antagonist IVF cycle using combination of Rekovelle and Menopur for stimulation according to the modified protocol employed at clinique ovo without deviation
* Presence of both ovaries

Exclusion Criteria:

* Second cycle of Duo-Stim IVF

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — in vitro fertilization can only be done on women as we have to stimulate ovaries
Study Population: Women consulting the clinic for fertility issues that require in vitro fertilization
Sampling Method: Non-Probability Sample
Enrollment: 772 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Identify the population where a simplified IVF monitoring is conceivable | Up to 3 weeks
  Rate of Rekovelle and / or Menopur dose modification before day 10 ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kadoch, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No